CLINICAL TRIAL: NCT06445569
Title: A Randomized, Double-blind, Placebo-controlled, Proof-of-concept Study to Evaluate the Safety and Efficacy of the Test Product KH-1 for Stimulating Autophagy in Non-diabetic Adults With Elevated Blood Glucose Concentration
Brief Title: Safety and Efficacy of KH-1 for Stimulating Autophagy in Non-diabetic Adults With Elevated Blood Glucose Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kalin Health, LLC (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: K02-21-01-T0012
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: PreDiabetes; Aging
Keywords: Elevated Blood Glucose; Spermidine; Autophagy; Probiotic
MeSH Terms: conditions — Prediabetic State; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Participants will consume their assigned study product for 3 months, after which all participants will be assigned to consume the KH-1 for the remaining 3 months in an open-label fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KH-1 (Active Comparator): Three capsules containing spermidine and amino acids. One stick packet containing probiotics.
  Interventions: Dietary Supplement: KH-1
- Placebo (Placebo Comparator): Three capsules containing hypromellose, hypromellose acetate succinate, purified water, pigments and gellen gum.
  One stick packet containing microcrystalline cellulose.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: KH-1 — 3 capsules and one stick packet consumed daily around the same time
  Arms: KH-1
Other: Placebo — 3 capsules and one stick packet consumed daily around the same time
  Arms: Placebo

SUMMARY:
Aging significantly impacts overall health and is a risk factor for developing diabetes. An estimated 50% of U.S. adults aged ≥65 years were reported to have prediabetes (defined as having a fasting glucose concentration of 100-125 mg/dl) in 2005-2008. The Centers for Disease Control and Prevention (CDC) has stated that in the United States, 88 million people (one in every 3 Americans) are currently classified as prediabetic, emphasizing the importance of preventative measures and early intervention to manage and reduce the risk of progression to diabetes. Additionally, an estimated 430 million individuals worldwide are expected to have prediabetes by 2030. Dietary supplementation of polyamines, spermidine in particular, have been touted to have beneficial health effects such as increasing life span and mitigating impacts of aging. Spermidine and spermine are polyamines that are being increasingly investigated for their ability to slow the aging process by inducing autophagy. Nevertheless, literature on these topics is scarce and results from trials have been inconclusive; therefore further research is needed. The novel nutraceutical KH-1, comprised of spermidine, spermidine derivatives and probiotics, is examined in this trial of healthy volunteers aged 18 years or over. This study evaluates KH-1 for its safety and its effect on glucose homeostasis. This study measures the effects of KH-1 on biomarkers for inflammation, cardiovascular disease, insulin sensitivity, and those important for autophagy. A qualitative assessment of the effect of KH-1 on well-being is also examined.

DETAILED DESCRIPTION:
Prediabetes is the intermediate state and precursor that can lead to an eventual diagnosis of diabetes. The presence of an elevated hemoglobin A1c (HbA1c), as well as insulin resistance with concomitant β-cell dysfunction is a strong indicator of prediabetes. Dietary and lifestyle changes are the most effective methods to control and prevent prediabetes, but maintenance of these changes is often difficult. Pharmaceutical options are indicated for treatment of diabetes rather than prevention of prediabetes, however many are associated with side effects. Therefore, a safe and effective alternative to prevent disease in metabolically dysregulated individuals is necessary.

The novel nutraceutical KH-1 is comprised of spermidine, amino acids, and a probiotic. This nutraceutical may offer a promising strategy for managing prediabetes.

This study is a double-blinded randomized controlled trial with 48 healthy volunteers to test the efficacy and safety of the novel nutraceutical KH-1. A total of 48 participants will be randomized in a double-blinded fashion, with 24 participants in each study group (KH-1 vs. placebo). After screening and randomization, participants will consume their assigned study product for 3 months, after which all participants will be assigned to consume the KH-1 for the remaining 3 months in an open-label fashion. Upon arrival at the clinic at the screening visit, participants will review the informed consent form (ICF), and if they agree to participate in the study, will sign and date the ICF, complete a brief screening, provide demographic information, and take part in other study activities indicated to be done on the screening visit. Participants who complete the screening process and qualify to continue are randomized to receive either the KH-1 or placebo in a 1:1 ratio for the first 3 months and assigned a unique randomization code. After the first 3 months, all participants will take KH-1. Participants will be instructed on the use of the nutraceutical product/placebo, according to label instructions. Participants will self-administer the study product at home and compliance will be assessed and documented at each visit. Venous blood samples will be collected at Week 0, Week 12 and Week 24 and analysed for biomarkers of glucose regulation and metabolism, cardiovascular health, inflammatory and autophagy biomarkers. Haematology and biochemistry parameters will be measured at screening, week 0, week 12 and week 24. A qualitative health questionnaire will be completed at 3 in-clinic visits and physical measurements to assess safety of the nutraceutical.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult participants who are at least 50 years of age (inclusive) at the time of signing the informed consent form.
2. Have a body mass index (BMI) between 25.0 to 45.0 kg/m2 (inclusive).
3. In good general health and good oral health (no active or uncontrolled diseases, infections or conditions).
4. Impaired glucose metabolism evidence by either fasting glucose of 100 to 125 mg/dL at screening or an HbA1c between 5.7 and 6.4%.
5. Female participants of childbearing potential (i.e., participants who are not surgically sterilized or not post-menopausal (defined as amenorrhea for greater than 1 year), or transgendered males with retained ovaries and uterus) must agree to use a medically approved method of birth control for at least one month prior (or three months prior in the case of oral or long-acting injective contraceptives) to the first dose of study product and throughout the study, or abstain from heterosexual intercourse throughout the duration of the study and have a negative urine pregnancy result at baseline. For males of reproductive potential: use of condoms, abstinence from heterosexual intercourse, or other methods to ensure that their partners (if able) do not become pregnant during the course of the study.
6. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion criteria:

1. Participant has a medical history of uncontrolled hypertension (i.e., ≥160 mmHg systolic and/or ≥100 mmHg diastolic)
2. Participant has a medical history of heart disease and/or cardiovascular disease, kidney disease (dialysis or renal failure), hepatic impairment or disease, or Type 1 or Type 2 diabetes.
3. Participant has a medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the year prior to screening, immune disorder (i.e., HIV/AIDS), or a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening visit.
4. Female participants who are lactating, pregnant, or planning to become pregnant during the study.
5. Have a known intolerance, sensitivity, or allergy to any of the study products or their ingredients, or any of the excipients used in the formulation.
6. Have a known intolerance, sensitivity, or allergy to milk.
7. Unable to be prescribed at least one of the antibiotics outlined in the study protocol.
8. Any condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the participant or the quality of the study data.
9. Currently taking dietary supplements other than vitamins (a 14-day washout period prior to baseline/Visit 2 would be permitted).
10. Taking any prescription medication at the time of randomization that is known to impact blood sugar and or blood sugar metabolism, as per Principal Investigator's (PI) discretion.
11. Use of certain medications in timeframes defined in the study protocol (Ampicillin, Gentamicin, Kanamycin, Streptomycin, Erythromycin, Clindamycin, Tetracycline, Chloramphenicol, Potassium sparing diuretics, Nitroglycerin and other nitrates, antidiabetic/Blood sugar lowering medications, any blood thinning medications (i.e., anticoagulant/antiplatelet drugs), antidepressants (use is permitted if dosage is maintained throughout the study), anxiolytics, antipsychotics , anticholinergics/antispasmodics, calcium-channel blockers (use is permitted if dosage is maintained throughout the study), Opioids.
12. Use of supplements dietary supplements/food/drink within 2 weeks or 7 half-lives (whichever is longer) prior to baseline and for the duration of the study, including foods/drinks rich in probiotics or prebiotics (e.g., yogurt, sauerkraut, kombucha) or synbiotics, Any herbs and supplements with hypoglycemic potential, any herbs or supplements that induce weight loss, any blood sugar lowering herbs or supplements, any blood thinning herbs or supplements
13. History of alcohol or substance abuse in the 12 months prior to screening.
14. Receipt or use of an investigational product in another research study within 28 days prior to baseline/Visit 2.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 3 months
  Between placebo and test product, change from baseline to 3 months in fasting insulin
Insulin resistance | 3 months
  Between placebo and test product, change from baseline to 3 months in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Insulin Resistance | 3 months
  Between placebo and test product, change from baseline to 3 months Oral Glucose Tolerance Test (OGTT)- derived indices of insulin dynamics

SECONDARY OUTCOMES:
Long-term effect on Insulin Resistance | 3 months
  Within-group change from baseline to 3 months for fasting insulin
Long-term effect on Insulin Resistance | 6 months
  Within-group change from baseline to 6 months for fasting insulin
Long-term effect on Insulin Resistance | 3 months
  Within-group change from baseline to 3 months for HOMA-IR
Long-term effect on Insulin Resistance | 6 months
  Within-group change from baseline to 6 months for HOMA-IR
Long-term effect on Insulin resistance | 3 months
  Within-group change from baseline to 3 months for OGTT-derived indices
Long-term effect on Insulin Resistance | 6 months
  Within-group change from baseline to 6 months for OGTT-derived indices
Post-prandial Glycemic Response | 3 months
  Between placebo and test product, change from baseline to 3 months in area under the glucose concentration (AUC) post-OGTT
Post-prandial Glycemic Response | 3 months
  Within-group change from baseline to 3 months in area under the glucose concentration (AUC) post-OGTT
Post-prandial Glycemic Response | 6 months
  Within-group change from baseline to 6 months in area under the glucose concentration (AUC) post-OGTT
Post-prandial Glycemic Response | 3 months
  Between placebo and test product, change from baseline to 3 months in 2-hour post-prandial glucose
Post-prandial Glycemic Response | 3 months
  Within-group change from baseline to 3 months in 2-hour post-prandial glucose
Post-prandial Glycemic Response | 6 months
  Within-group change from baseline to 6 months in 2-hour post-prandial glucose
Glycemic Control | 3 months
  Between placebo and test product, change from baseline to 3 months in fasting glucose
Glycemic Control | 3 months
  Within-group change from baseline to 3 months in fasting glucose
Glycemic Control | 6 months
  Within-group change from baseline to 6 months in fasting glucose
Glycemic Control | 3 months
  Between placebo and test product, change from baseline to 3 months in HbA1c
Glycemic Control | 3 months
  Within-group change from baseline to 3 months in HbA1c
Glycemic Control | 6 months
  Within-group change from baseline to 6 months in HbA1c
β-cell Function | 3 months
  Between placebo and test product, change from baseline to 3 months in oral disposition index (DI) calculated by the ratio of the insulinogenic index over fasting insulin
β-cell Function | 3 months
  Within-group change from baseline to 3 months in oral DI
β-cell Function | 6 months
  Within-group change from baseline to 6 months in oral DI
Cardiovascular Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in fasting triglycerides (TG)
Cardiovascular Biomarkers | 3 months
  Within-group change from baseline to 3 months in fasting TG
Cardiovascular Biomarkers | 6 months
  Within-group change from baseline to 6 months in fasting TG
Cardiovascular Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in fasting total cholesterol
Cardiovascular Biomarkers | 3 months
  Within-group change from baseline to 3 months in fasting total cholesterol
Cardiovascular Biomarkers | 6 months
  Within-group change from baseline to 6 months in fasting total cholesterol
Cardiovascular Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in fasting low-density lipoprotein (LDL)
Cardiovascular Biomarkers | 3 months
  Within-group change from baseline to 3 months in fasting LDL
Cardiovascular Biomarkers | 6 months
  Within-group change from baseline to 6 months in fasting LDL
Cardiovascular Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in high-density lipoprotein (HDL)
Cardiovascular Biomarkers | 3 months
  Within-group change from baseline to 3 months in HDL
Cardiovascular Biomarkers | 6 months
  Within-group change from baseline to 6 months in HDL
Inflammatory Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in high-sensitivity C-reactive protein (hs-CRP)
Inflammatory Biomarkers | 3 months
  Within-group change from baseline to 3 months in hs-CRP
Inflammatory Biomarkers | 6 months
  Within-group change from baseline to 6 months in hs-CRP
Inflammatory Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in tumor necrosis factor (TNF)-alpha
Inflammatory Biomarkers | 3 months
  Within-group change from baseline to 3 months in TNF-alpha
Inflammatory Biomarkers | 6 months
  Within-group change from baseline to 6 months in TNF-alpha
Inflammatory Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in interleukin-6 (IL-6)
Inflammatory Biomarkers | 3 months
  Within-group change from baseline to 3 months in IL-6
Inflammatory Biomarkers | 6 months
  Within-group change from baseline to 6 months in IL-6
Autophagy | 3 months
  Between placebo and test product, change from baseline to 3 months in Beclin-1
Autophagy | 3 months
  Within-group change from baseline to 3 months in Beclin-1
Autophagy | 6 months
  Within-group change from baseline to 6 months in Beclin-1
Immunity Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in Cluster of Differentiation (CD) 3
Immunity Biomarkers | 3 months
  Within-group change from baseline to 3 months in CD3
Immunity Biomarkers | 6 months
  Within-group change from baseline to 6 months in CD3
Immunity Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in CD4
Immunity Biomarkers | 3 months
  Within-group change from baseline to 3 months in CD4
Immunity Biomarkers | 6 months
  Within-group change from baseline to 6 months in CD4
Immunity Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in CD8
Immunity Biomarkers | 3 months
  Within-group change from baseline to 3 months in CD8
Immunity Biomarkers | 6 months
  Within-group change from baseline to 6 months in CD8
Immunity Biomarkers | 3 months
  Between placebo and test product, change from baseline to 3 months in CD25
Immunity Biomarkers | 3 months
  Within-group change from baseline to 3 months in CD25
Immunity Biomarkers | 6 months
  Within-group change from baseline to 6 months in CD25
Overall Patient Health | 3 months
  Between placebo and test product, change from baseline to 3 months in Patient Health Questionnaire scores
Overall Patient Health | 3 months
  Within-group change from baseline to 3 months in Patient Health Questionnaire scores
Overall Patient Health | 6 months
  Within-group change from baseline to 6 months in Patient Health Questionnaire scores
Overall Quality of Life | 3 months
  Between placebo and test product, change from baseline to 3 months in RAND-36 questionnaire scores
Overall Quality of Life | 3 months
  Within-group change from baseline to 3 months in RAND-36 questionnaire scores
Overall Quality of Life | 6 months
  Within-group change from baseline to 6 months in RAND-36 questionnaire scores
Stress | 3 months
  Between placebo and test product, change from baseline to 3 months in Perceived Stress Scale (PSS) scores
Stress | 3 months
  Within-group change from baseline to 3 months in PSS scores
Stress | 6 months
  Within-group change from baseline to 6 months in PSS scores
Systolic Blood Pressure (SBP) | 6 months
  Change from baseline to 6 months in SBP (mmHg)
Diastolic Blood Pressure (DBP) | 6 months
  Change from baseline to 6 months in DBP (mmHg)
Heart Rate | 6 months
  Change from baseline to 6 months in heart rate (beats per minute)
Weight | 6 months
  Change from baseline to 6 months in weight (kg)
Percent Body Fat | 6 months
  Change from baseline to 6 months in percent body fat (%)
Body Mass Index (BMI) | 6 months
  Change from baseline to 6 months in BMI (kg/m2)
Whole Blood Hemoglobin | 6 months
  Change from baseline in fasting whole blood hemoglobin (g/dL)
Whole Blood Hematocrit | 6 months
  Change from baseline in fasting whole blood hematocrit (%)
Whole Blood Red Blood Cell Count | 6 months
  Change from baseline in fasting whole blood red blood cell count (x10^6/uL)
Whole Blood Red Blood Cell Distribution Width | 6 months
  Change from baseline in fasting whole blood red blood cell distribution width (%)
Whole Blood Mean Corpuscular Volume | 6 months
  Change from baseline in fasting whole blood mean corpuscular volume (fL)
Whole Blood Mean Corpuscular Hemoglobin | 6 months
  Change from baseline in fasting whole blood mean corpuscular hemoglobin (pg)
Whole Blood Mean Corpuscular Hemoglobin Concentration | 6 months
  Change from baseline in fasting whole blood mean corpuscular hemoglobin concentration (g/dL)
Whole Blood White Blood Cells | 6 months
  Change from baseline in fasting whole blood white blood cells (x10^3/uL)
Whole Blood Neutrophils | 6 months
  Change from baseline in fasting whole blood neutrophils (cells/uL)
Whole Blood Basophils | 6 months
  Change from baseline in fasting whole blood basophils (cells/uL)
Whole Blood Eosinophils | 6 months
  Change from baseline in fasting whole blood eosinophils (cells/uL)
Whole Blood Lymphocytes | 6 months
  Change from baseline in fasting whole blood lymphocytes (cells/uL)
Whole Blood Monocytes | 6 months
  Change from baseline in fasting whole blood monocytes (cells/uL)
Whole Blood Mean Platelet Volume | 6 months
  Change from baseline in fasting whole blood mean platelet volume (fL)
Whole Blood Platelet Count | 6 months
  Change from baseline in fasting whole blood platelet count (x10^9/L)
Serum Creatinine | 6 months
  Change from baseline in fasting serum creatinine (umol/L)
Serum Blood Urea Nitrogen | 6 months
  Change from baseline in fasting serum blood urea nitrogen (mg/dL)
Serum Alkaline Phosphatase (ALP) | 6 months
  Change from baseline in fasting serum ALP (U/L)
Serum Asparatate Transaminase (AST) | 6 months
  Change from baseline in fasting serum AST (U/L)
Serum Alanine Transaminase (ALT) | 6 months
  Change from baseline in fasting serum ALT (U/L)
Serum Albumin | 6 months
  Change from baseline in fasting serum albumin (g/dL)
Serum Total Protein | 6 months
  Change from baseline in fasting serum total protein (g/dL)
Serum Chloride | 6 months
  Change from baseline in fasting serum chloride (mmol/L)
Serum Sodium | 6 months
  Change from baseline in fasting serum sodium (mmol/L)
Serum Potassium | 6 months
  Change from baseline in fasting serum potassium (mmol/L)
Serum Calcium | 6 months
  Change from baseline in fasting serum calcium (mg/dL)
Serum Urea | 6 months
  Change from baseline in fasting serum urea (mg/dL)
Incidence of Adverse Events | 6 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Velasquez, MD, Principal Investigator — LifeDOC Research, PLLC
Locations (1):
- LifeDOC Research, PLLC, Memphis, Tennessee, United States